CLINICAL TRIAL: NCT06167434
Title: Clinical Investigation of the Future Cardia™ Insertable Cardiac Monitor in Subjects With Paroxysmal Atrial Fibrillation Voice Of the Heart Trial (First-in-Human Study)
Brief Title: Future Cardia™ Insertable Cardiac Monitor in Subjects With Paroxysmal Atrial Fibrillation (First-in-Human Study)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future Cardia, Inc (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FC-2022-01
Record Dates: First submitted 2023-11-21; First posted 2023-12-12 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-03

CONDITIONS: Arrhythmias, Cardiac; Atrial Fibrillation; Bradycardia; Ventricular Tachycardia; Asystole
Keywords: Telemedicine; Cardiac Arrhythmia; ECG; PCG; Accelerometer; Cardiac monitor; Insertable cardiac monitor
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Bradycardia; Tachycardia, Ventricular; Heart Arrest | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Experimental): Insertable Cardiac Monitor Implant.
  Interventions: Device: Future Cardia™ Insertable Cardiac Monitoring (ICM) System

INTERVENTIONS:
Device: Future Cardia™ Insertable Cardiac Monitoring (ICM) System — The Future Cardia™ ICM procedure will be performed as a stand-alone procedure for subcutaneous insertion.

SUMMARY:
This study is a first-in-human, prospective, multi-center, pre-market single-arm clinical trial to evaluate the Future Cardia™ ICM.

DETAILED DESCRIPTION:
The objective of this first-in-human, prospective, multi-center, pre-market single-arm clinical investigation is to evaluate the safety and performance of the Future Cardia™ ICM by assessing the insertion procedure, sensing and detection performance and data monitoring transmission success, and device- or procedure-related complication rates over a 6-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years old and <75 years old)
2. Paroxysmal AF, defined as AF that terminates spontaneously or with intervention within 7 days of onset (ESC 2020 guidelines). In order to be included, patients must present one of the following conditions:

   1. paroxysmal AF patients that are candidates for AF ablation;
   2. patients hospitalized for symptomatic AF, who failed to convert in the emergency room (ER):
   3. outpatients who require treatment with anti-arrhythmic drugs (AAD) (mostly propafenone or flecainide; more rarely sotalol or amiodaron are given for PAF).
3. Patient is willing and able to provide written informed consent.
4. Patient is willing and able to comply with the protocol, including follow-up visits and data transmissions.

Exclusion Criteria:

1. Patient who is scheduled to have MRI or is likely to require MR screening. The Future Cardia implant is not compatible with MRI.
2. Currently indicated for or implanted with a cardiovascular implantable electronic device (CIED) (e.g., ICM or ILR, pacemaker, ICD, CRT-D or CRT-P device) or hemodynamic monitoring system.
3. Compromised immune system or at high risk of developing an infection.
4. Active systemic infection or history of any infection within the last 30 days.
5. Subjects who are female must:

   1. have a negative pregnancy test by β-hCG blood test.
   2. not breastfeeding
   3. either be surgically sterile, postmenopausal (cessation of menses for at least 1 year), or if they have childbearing potential, agree to use a medically accepted, highly effective method of contraception during the entire duration of the study.
6. Subject is currently enrolled in another investigational study.
7. Any condition or abnormality (including clinical laboratory, physical examination, or vital sign abnormalities), current or past, that, in the opinion of the Investigator, would compromise the efficacy evaluation, safety of the patient, or would interfere with or complicate study procedures or assessments.
8. Any concomitant condition which, in the opinion of the investigator, would not allow safe participation in the study (e.g., drug addiction, alcohol abuse, emotional/psychological diagnosis).
9. Obesity, Class 2 (BMI ≥ 35-40) or Class 3 (BMI ≥ 40).
10. Subject is unwilling or unable to comply with the study procedures.
11. Subject is legally incapacitated and unable to provide written informed consent.

    Exclusion criteria for the study procedure:
12. Patient with abnormal thoracic anatomy or scar tissue at the implant site that may adversely impact the insertion procedure.
13. For patients currently taking warfarin at the time of insertion, most recent INR value (within 7 days) is less than 3.5 for an acceptable risk of bleeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of Insertion Procedure - Implantation: Insertion Success | up to 24 weeks
  Insertion Success. (Yes/No); Place Device into Pocket (Yes/No);
Characterization of Insertion Procedure - Implantation: Incision Size | up to 24 weeks
  Incision Size in millimeters (mm).
Characterization of Insertion Procedure - Implantation: Device Orientation | up to 24 weeks
  Device Orientation: Location between the suprasternal notch and the left nipple, (position A); or left parasternal region (position B) or left sub-mammary position can be used (position C).
Characterization of Insertion Procedure - Implantation: Duration of Insertion Procedure. | up to 24 weeks
  Duration of Insertion Procedure in minutes (min).
Characterization of Explant Procedure - Device removal: Removal Success | up to 24 weeks
  Removal Success (Yes/No)
Characterization of Explant Procedure - Device removal: Incision Size | up to 24 weeks
  Incision Size in millimeters (mm)
Characterization of Explant Procedure - Device removal: Duration of explant procedure | up to 24 weeks
  Duration of explant procedure in minutes (min).
Device and Procedural Safety over a period of 180 days | up to 24 weeks
  1. Number of Serious Adverse Events (SAE) related to the Device or insertion procedure.
  2. Number of Participants with Device-related or Procedure-related Serious Adverse Event that require additional invasive intervention (including need to for device removal, device replacement, surgical repositioning of the device, or another surgery related to the device or primary insertion procedure).
Success of Wireless Transmissions over a period of 180 days | up to 24 weeks
  Assess the percentage of successful wireless transmissions from the system throughout the study duration (transmission successful, the transmission failed or transmission re-try).

SECONDARY OUTCOMES:
Evaluation of the sensing quality of Future Cardia™ ICM, through assessment of the ECG signal by two independent electrophysiologists. | up to 24 weeks
  ECG signal Assessment.
Comparison of the Future Cardia™ ECG tracing and detection of arrhythmias with 7-day ECG recorder tracings or 24-hr Holter recording (optional, when available). | up to 24 weeks
  Comparison of the Future Cardia™ ECG tracing and detection of arrhythmias with 7-day ECG recorder tracings or 24-hr Holter recording.
Usability: survey of the implanting physicians regarding the ease of implantation and use of the system for monitoring during follow-up. | up to 24 weeks
  Usability Survey
Number of Serious Adverse Events (SAE) related to the Device or study procedure in patients who elect to continue monitoring using the ICM device after the 6-month study follow-up. | 2 Years
  Long-term safety in Post study follow-up (> 6 months up to 2 years).

CONTACTS AND LOCATIONS:
Overall Officials: Ante Anic, MD, Principal Investigator — University Hospital of Split
Locations (1):
- University Hospital of Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Future Cardia Inc.Website — https://futurecardia.com/
- See also: Meditrial Europe Ltd.CRO — https://www.meditrial.net/